CLINICAL TRIAL: NCT01635257
Title: Accuracy of Multi-organ Ultrasound (Venous, Cardiac and Thoracic) for the Diagnosis of Pulmonary Embolism: Suspected Pulmonary Embolism Sonographic Assessment (SPES) Multicenter Prospective Study
Brief Title: Accuracy of Multi-organ Ultrasound for the Diagnosis of Pulmonary Embolism
Acronym: SPES
Status: Completed | Type: Observational
Sponsor: Azienda Ospedaliero-Universitaria Careggi (Other)
Responsible Party: Principal Investigator, Peiman Nazerian, Medical Doctor Emergency Medicine, Azienda Ospedaliero-Universitaria Careggi
Other Study IDs: 080974
Record Dates: First submitted 2012-07-01; First posted 2012-07-09 (Estimated); Last update posted 2013-03-18 (Estimated); Status verified 2013-03

CONDITIONS: Pulmonary Embolism
Keywords: pulmonary embolism diagnosis; ultrasound
MeSH Terms: conditions — Pulmonary Embolism | interventions — High-Energy Shock Waves

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- suspected pulmonary embolism patients: patients with clinical suspicion of PE and with a simplified Well's score>4 (PE likely) or with a D-dimer value ≥500ng/ml presenting to the emergency departments of Careggi University Hospital (Firenze), of San Luigi Gonzaga University Hospital (Torino) of Ospedale Pierantoni-Morgagni (Forlì)
  Interventions: Other: Ultrasound scan

INTERVENTIONS:
Other: Ultrasound scan — A multiorgan ultrasound was performed by an emergency physician sonographer before MCTPA. Pulmonary embolism was considered echographically present if compression ultrasound was positive for deep vein thrombosis or transthoracic-echocardiography was positive for right ventricular dysfunction or at least one pulmonary subpleural infarct was detected with thoracic ultrasound.

SUMMARY:
Patients with suspected Pulmonary Embolism (PE) and a high clinical probability or a high D-dimer level should undergo a second level diagnostic test such as Multidetector Computed Tomography Angiography (MCTPA). Unfortunately MCTPA involves radiation exposure, is expensive, is not feasible in unstable patients and has contraindications. UltraSound (US) is safe and rapidly available even in unstable patients. Many authors evaluated the diagnostic role of Compression Ultrasound Scan (CUS) for detecting limbs Deep Vein Thrombosis (DVT), TransThoracic Echocardiography (TTE) for detecting Right Ventricular Dysfunction (RVD) or Thoracic UltraSound (TUS) for detecting subpleural infarcts in patients with suspected PE. No previous studies have investigated the diagnostic accuracy of CUS, TTE and TUS combined (multiorgan US) for the diagnosis of PE. This study evaluates the diagnostic accuracy of multiorgan US.

Methods. Consecutive patients that underwent MCTPA in the Emergency Department for clinical suspicion of PE and with a simplified Well's score>4 (PE likely) or with a D-dimer value ≥500ng/ml were enrolled in the study. MCTPA was considered the gold standard for PE diagnosis. A multiorgan US was performed by an emergency physician sonographer before MCTPA. PE was considered echographically present if CUS was positive for DVT or TTE was positive for RVD or at least one pulmonary subpleural infarct was detected with TUS. The accuracy of the single and multiorgan US was calculated.

ELIGIBILITY:
Inclusion Criteria:

* Patients with clinical suspected pulmonary embolism
* Simplified Well's score>4 (PE likely) or D-dimer value ≥500ng/ml
* Patients that undergo MCTPA in the Emergency Department for suspected pulmonary embolism

Exclusion Criteria:

* Refused consent
* Less than 18 years old
* Not possible to perform ultrasound scan within 3 hours before MCTPA

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients more than 18 years presenting to three emergency departments with clinical suspected pulmonary embolism. Clinical suspected pulmonary embolism is defined as new onset or worsening dyspnea, chest pain, syncope or shock/Hypotension without an alternative obvious cause
Sampling Method: Non-Probability Sample
Enrollment: 357 (Actual)
Dates: Start 2012-06; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Accuracy of ultrasound for the diagnosis of pulmonary embolism | The goldstandard for PE diagnosis is the MCTPA performed within 24 hours from ED presentation. The recruiting period is 5 months. There is not a follow-up for the included patients.
  Sensitivity, specificity, negative and positive predictive value, negative and positive likelihood ratio of limb, cardiac, thoracic and multi-organ ultrasound for the diagnosis of pulmonary embolism in the emergency department considering as gold standard the Multidetector Computed Tomography Angiography (MCTPA)

CONTACTS AND LOCATIONS:
Overall Officials: Stefano Grifoni, MD, Study Chair — Director of Pronto Soccorso generale of AUO Careggi
Locations (3):
- Italy (3):
  - Emergency Department Azienda Ospedaliera Universitaria Careggi, Florence, Tuscany
  - Department of Emergency Medicine, Pierantoni Morgagni Hospital, Forlì
  - Department of Emergency Medicine, San Luigi Gonzaga University Hospital, Torino

REFERENCES:
- [Derived] Nazerian P, Vanni S, Volpicelli G, Gigli C, Zanobetti M, Bartolucci M, Ciavattone A, Lamorte A, Veltri A, Fabbri A, Grifoni S. Accuracy of point-of-care multiorgan ultrasonography for the diagnosis of pulmonary embolism. Chest. 2014 May;145(5):950-957. doi: 10.1378/chest.13-1087. PMID 24092475